CLINICAL TRIAL: NCT03268031
Title: Development of Artificial Intelligence-assissted Diagnostic Program of Glaucoma
Brief Title: Artificial Intelligence-assissted Glaucoma Evaluation
Acronym: AGE
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Xiulan Zhang, Director of Clinical Research Center, Sun Yat-sen University
Other Study IDs: ProjectAGE
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Artificial Intelligence; Glaucoma
Keywords: artificial intelligence; glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Visual Fields

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Glaucoma patients: Glaucoma patients will take visual field test and OCT imaging of optic nerve area. All of these data will be collected as source of machine learning.
  Interventions: Diagnostic Test: Visual field and OCT tests
- Non-glaucoma participants: Non-glaucoma participants will take visual field test and OCT imaging of optic nerve area. All of these data will be collected as source of machine learning.
  Interventions: Diagnostic Test: Visual field and OCT tests

INTERVENTIONS:
Diagnostic Test: Visual field and OCT tests — Visual field test and OCT are commonly used essential tests to make accurate diagnosis of glaucoma. Algorithms to classify Visual field and OCT tests would both be developed and verified.

SUMMARY:
Glaucoma is currently the second leading cause of irreversible blindness in the world. Our study intends to combine clinical data of glaucoma patients in Zhongshan Ophthalmic Center with Artificial Intelligence techniques to create programs that can screen and diagnose glaucoma.

DETAILED DESCRIPTION:
Glaucoma is currently the second leading cause of irreversible blindness in the world, which brings heavy burden to human society. Compared to other ocular diseases, diagnostic process of glaucoma is complicated depends on multiple test results, including visual field test, OCT, etc. How to diagnose glaucoma correctly and fast has always been a hot topic in glaucoma researches. Artificial intelligence is used to study and develop theories and methods that can help simulate and extend human intelligence, which has been utilized in a lot of research fields such as automatic drive and medicine. The study intends to combine clinical data of glaucoma patients in Zhongshan Ophthalmic Center with Artificial Intelligence techniques to create programs that can screen and diagnose glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. BCVA>0.1
2. able to complete reliable visual field test
3. no history of intraocular surgery or fundus laser

Exclusion Criteria:

1. unable to complete visual field test

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anyone who can complete visual field test and have BCVA>0.1 can be enrolled. We will collect visual field test result and OCT images of both glaucoma and non-glaucoma patients.
Sampling Method: Non-Probability Sample
Enrollment: 10800 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of diagnosis by artificial intelligence algorithm | from August 2017 to February 2021
  Accuracy of diagnosis by artificial intelligence algorithm and compare this result with glaucoma specialists

SECONDARY OUTCOMES:
Sensitivity of diagnosis by artificial intelligence algorithm | from August 2017 to February 2021
  Sensitivity of diagnosis by artificial intelligence algorithm
Specificity of diagnosis by artificial intelligence algorithm | from August 2017 to February 2021
  Specificity of diagnosis by artificial intelligence algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Xiulan Zhang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Diprose W, Buist N. Artificial intelligence in medicine: humans need not apply? N Z Med J. 2016 May 6;129(1434):73-6. PMID 27349266
- [Result] Quigley HA. Glaucoma. Lancet. 2011 Apr 16;377(9774):1367-77. doi: 10.1016/S0140-6736(10)61423-7. Epub 2011 Mar 30. PMID 21453963
- [Result] Asaoka R, Murata H, Iwase A, Araie M. Detecting Preperimetric Glaucoma with Standard Automated Perimetry Using a Deep Learning Classifier. Ophthalmology. 2016 Sep;123(9):1974-80. doi: 10.1016/j.ophtha.2016.05.029. Epub 2016 Jul 7. PMID 27395766